CLINICAL TRIAL: NCT04888078
Title: Incidence of POUR in the Veteran Population After Elective Inguinal Hernia Repair: A Retrospective Study
Brief Title: Bassini Inguinal Hernia Repair: Obsolete Or Still A Viable Surgical Option?
Status: Completed | Type: Observational
Sponsor: Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jeannie Rivers, Chief of Surgery, Hunter Holmes Mcguire Veteran Affairs Medical Center
Other Study IDs: 02331
Record Dates: First submitted 2021-05-11; First posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Inguinal Hernia; Surgery--Complications; Surgical Complication
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Bassini hernia repair — Non-mesh tissue inguinal hernia repairs

SUMMARY:
Retrospective review of hernia surgery patients at HHMcGuire VAMC focusing on repair type and postoperative complications.

ELIGIBILITY:
Inclusion Criteria: Inguinal hernia repair without mesh -

Exclusion Criteria: Mesh repair

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Veterans who underwent inguinal hernia repair without mesh
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Inguinal hernia recurrence | 5-13 years postoperatively
  chart review

SECONDARY OUTCOMES:
wound infection | 5-13 years
  chart review
urinary retention | 5-13 years
  chart review
groin pain | 5-13 years
  chart review
durability of repair | 5-13 years postop
  chart review
testicular ischemia | 5-13 years
  chart review

CONTACTS AND LOCATIONS:
Locations (1):
- Hunter Holmes McGuire VAMC, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
All personally identifiable information is secured. Study outcomes reported in aggregate only.